CLINICAL TRIAL: NCT05747872
Title: Effectiveness of Buerger Allen Exercise on Lower Extremity Perfusion and Wound Healing Among Type 2 Diabetes Mellitus Patients With Foot Ulcer: A Randomized Controlled Trial
Brief Title: Effectiveness of Buerger Allen Exercise Among Type 2 Diabetes Mellitus Patients With Foot Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Naile Bilgili, Professor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2021 - 814
Record Dates: First submitted 2023-01-19; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention Grup (Experimental): Buerger Allen exercises programme will be applied to the type 2 diabetes mellitus patients with foot ulcer. Patients in the intervention group performed daily Buerger Allen exercises for 12 weeks. Patients in the study intervention group were taught Buerger Allen exercises and were asked to exercise twice daily for 12 weeks. Individuals will be given an exercise diary, including the pictures of the exercises, to better manage this process. Reminder phone calls were made once a week to support the exercise program and increase motivation.
  Interventions: Behavioral: Buerger Allen Exercises
- Control Grup (No Intervention): The control group received standard wound care but no exercises.

INTERVENTIONS:
Behavioral: Buerger Allen Exercises — These exercises are specific exercises aimed at improving circulation in the feet and legs.
  While doing the exercises, first of all;
  1. The legs are raised at an angle of 45 degrees and supported in this position for 1-3 minutes until the skin turns white.
  2. Sit on the edge of the bed and let your legs hang down (make sure there is no pressure behind the knees). In this position, move your foot left and right and up and down for 3 minutes.
  3. Lie on your back for 5 minutes keeping your legs warm with a blanket.
  Performing all three of these exercises in sequence means 1 session. Exercises are done 2 times a day, at least 3 sessions each time.
  Arms: İntervention Grup

SUMMARY:
This study was conducted to determine the effect of Buerger Allen exercises on lower extremity perfusion and wound healing in patients with foot ulcer type 2 diabetes. The Buerger Allen exercise is a specific exercise that aims to improve circulation in the feet and legs. Buerger Allen exercise is an ideal and noninvasive therapy for diabetic patients with a diabetic foot ulcer as it is an easy-to-learn, repetitive, low-cost, and low-risk physical activity. Subjects were randomly allocated to either the control or intervention group. The ulcers and lower extremity perfusion of the patients in both the intervention and control groups were examined and measured.

DETAILED DESCRIPTION:
The purpose of this study was to investigate the effect of Buerger Allen exercises on lower extremity perfusion and wound healing in type 2 diabetic patients with a diabetic foot ulcer. Subjects were recruited by the researcher in the clinics where they received treatment. Randomized controlled study design was used in the study. Patients in the study were allocated to the control and study intervention groups. The data collection form developed by the researcher was used to collect the data. Patients in both groups received standard wound care. Subjects in the study intervention group were asked to exercise twice daily for 12 weeks. The ulcers and lower extremity perfusion of the groups were assessed in the beginning, in the 4th week, and the 12th week. The groups will be compared in terms of the ulcer size and lower extremity perfusion.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older,
* Patients with type 2 diabetes with foot ulcer
* Receiving oral antidiabetic and/or insulin therapy,
* PEDIS Classification stage 1 and 2
* Does not have communication and mental problems,
* are literate and speak Turkish,
* Patients who volunteered to participate in the study

Exclusion Criteria:

* with dementia and mental problems,
* Those with serious diabetes complications such as kidney failure and hemodialysis,
* Patients receiving hyperbaric oxygen therapy, negative pressure wound therapy, epidermal growth factor for wound healing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-10-17 (Actual)

PRIMARY OUTCOMES:
Change in Ankle Brachial Index (ABI) | Change from baseline Ankle Brachial İndex (ABI) at 12 weeks
  To calculate the ABI, each ankle systolic pressure was divided by the brachial systolic pressure and the higher of the two systolic pressures for each leg was divided by the higher of the two arm pressures to get the right and left ABI The score was interpreted as
  * above 0.9 (normal perfusion),
  * 0.71-0.90 (mildly impaired perfusion),
  * 0.41-0.70 (moderately impaired perfusion),
  * below 0.40 (severely impaired perfusion).
Change in ulcer surface area | Change from baseline ulcer surface area at 12 weeks
  Ulcer size was measured in centimeters. Ulcer surface area was measured using a scaled transparent measurement paper.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Çankaya, Turkey (Türkiye)